CLINICAL TRIAL: NCT00889200
Title: Eszopiclone Treatment & Cortisol Response to HPA Axis Tests
Brief Title: Eszopiclone Treatment & Cortisol Responsivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0608-002
Record Dates: First submitted 2009-04-23; First posted 2009-04-28 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label Eszopiclone (Experimental): Standard dosing of drug for 6 weeks for insomnia
  Interventions: Drug: eszopiclone

INTERVENTIONS:
Drug: eszopiclone — 6 weeks standard oral therapy
  Other Names: Lunesta

SUMMARY:
This study was designed to use a sensitive neuroendocrine probe, the Dexamethasone/Corticotropin-Releasing Hormone (DEX/CRH) test, in a sample of healthy adults with insomnia. The primary aim was to assess cortisol reactivity before and after long-term (6 weeks) administration of eszopiclone. It was hypothesized that treatment with eszopiclone would result in a significant reduction in plasma cortisol response to the DEX/CRH test following treatment of insomnia with standard dose of eszopiclone.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate Insomnia

Exclusion Criteria:

* Any acute or chronic medical condition involving function of HPA axis (e.g., Cushing's or Addison's Disease, adrenal or pituitary gland disorders)
* Currently taking, or unable to be free of, antidepressant, neuroleptic, anxiolytic, or thymoleptic drugs for at least 2 weeks preceding the DEX/CRH test (free of fluoxetine for at least 6 weeks)
* Current use of psychotropic medication or medication (prescribed or over the counter) thought to affect HPA axis function or glucocorticoid synthesis/release (e.g., prednisone, anabolic steroids, DHEA, ketoconazole, metyrapone)
* History of a significant adverse reaction to eszopiclone
* Meets DSM-IV criteria for any Axis I psychiatric disorder, including substance abuse presently, or substance dependence within the past 6 months
* Pregnancy, lactation, or unable/unwilling to use reliable methods of contraception during the study procedures
* Limited mental competency and the inability to give informed, voluntary, written consent to participate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Carpenter, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the community via flyers and through Internet and newspaper advertisements for "healthy adults experiencing problems with sleep." Voluntary written informed consent was obtained for the study, which was approved by the Butler Hospital Institutional Review Board.
Pre-assignment Details: Excluded subjects met criteria for current major depressive disorder (MDD) or other major Axis I psychiatric or substance use disorders. Subjects reporting < 6 hours of sleep/night and with score > 10 on Insomnia Severity Index (ISI) qualified. General good health required on physical and neurological examinations and on laboratory studies.
Groups:
- Open-label Eszopiclone: Standard daily dosing of 3 mg drug nightly for 6 weeks for insomnia
  eszopiclone : 6 weeks standard oral therapy
Period: Overall Study
Arm/Group | Open-label Eszopiclone
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-label Eszopiclone: Standard dosing of drug for 6 weeks for insomnia
  eszopiclone : 6 weeks standard oral therapy
Arm/Group | Open-label Eszopiclone
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Depressive Symptoms [Mean (Standard Deviation); unit: scores on a scale] — Inventory for Depressive Symptomology-Self Report version (IDS-SR), total score calculated without 4 items pertaining to sleep. Range of scores on this version of the IDSSR are 0 (best outcome; no symptoms) to 69 (worst outcome; severe symptoms).
  scores on a scale | 13.83 (8.24)
plasma cortisol response to standardized dexamethasone/Corticotropin Releasing Hormone (DEX/CRH) [Mean (Standard Deviation); unit: nmol/L] — Cortisol assays were performed on plasma samples from 2:59 PM (baseline), 3:30 PM, 3:45 PM, 4:00 PM, 4:15 PM, and 5:00 PM. Radioimmunoassay (RIA) used to measure cortisol in duplicate at each time point; intra-assay and inter-assay coefficients of variation observed for quality assessment samples (5 and 20 nmol/L) were <5% and 10%, respectively. Cortisol "response"was summarized by absolute change from pre-CRH infusion (time point 0) to peak level after CRH infusion.
  nmol/L | 146.23 (161.85)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Self report measure of Insomnia. Subjects had to have a total score >10 to enroll. The range of the scales is from 0 (no insomnia symptoms) to 28 (severe insomnia symptoms).
  units on a scale | 15.23 (2.93)

OUTCOME MEASURES:

1. Primary Outcome: Cortisol Response to the Dex/CRH Test Post-treatment (6 Weeks Oral Drug)
Description: Cortisol reponse to the DEX/CRH test post-treatment is the same as measured and calculated at baseline =delta(CORT).
Time Frame: post drug (6 weeks oral eszopiclone)
Population: All subjects completed all study procedures
Measure: Mean (Standard Deviation); unit: nmol/L
Units Other Than Participants: paired t-test cortisol reactivity
Groups:
- Open-label Eszopiclone: After Standard dosing of drug for 6 weeks for insomnia, Dex/CRH test was repeated to measure cortisol reactivity with the same neuroendocrine test
Arm/Group | Open-label Eszopiclone
Number analyzed (Participants) | 12
Number analyzed (paired t-test cortisol reactivity) | 12
nmol/L | 108.98 (129.19)

ADVERSE EVENTS:
Time Frame: Over 6 weeks on drug; verbal report by subject at clinic assessments every 2 weeks
Arm/Group | Open-label Eszopiclone
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No